## **COVER PAGE**

## STATISTICAL ANALYSIS PLAN

**OFFICIAL TITLE:** The Effects of Motivational Messages Sent to Emergency Nurses during the COVID-19 Pandemic on Job Satisfaction, Compassion Fatigue, and Communication Skills: A Randomized Controlled Trial

**DATE OF DOCUMENT**: May 06, 2021

## Statistical Analysis Plan

The study data were analyzed using SPSS for Windows version 22.0 (IBM Corp, Armonk, NY). Number, percentage, mean, and standard deviation were used as descriptive statistical methods The normal distribution was evaluated with kurtosis and skewness. The distribution of descriptive features according to the groups was tested by chi-square analysis. For comparison of quantitative continuous data between two independent groups, t-test, within-group changes were analyzed by Repeated Measures ANOVA test. A p value of < .05 was considered statistically significant.